CLINICAL TRIAL: NCT00057148
Title: Acute Post-Operative Pain Management Using Massage As Adjuvant Therapy
Brief Title: Massage After Surgery To Help Treat Post-Operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 01-197
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-03

CONDITIONS: Postoperative Pain
Keywords: massage therapy; pain management; post-surgical; complementary therapy
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: massage treatment

INTERVENTIONS:
Procedure: massage treatment

SUMMARY:
Postoperative pain is often undertreated. Although studies have demonstrated that many patients experience a substantial degree of unrelieved pain following operative procedures and that this pain can increase the incidence of serious complications, the management of discomfort continues to be suboptimal. Narcotic analgesia is the mainstay of acute postoperative pain management but patient, clinician, and institutional barriers often limit the effectiveness of drug treatment. Furthermore, pharmacologic interventions alone may not address all the factors involved in the conscious experience of pain. Massage is a complementary or adjunctive medical technique that has been used for thousands of years. Yet there is scant research related to the use of massage therapy in postoperative pain management. Used in tandem with pharmacologic treatments, massage may have the potential to substantially improve acute pain relief.

DETAILED DESCRIPTION:
BACKGROUND / RATIONALE:

Postoperative pain is often undertreated. Although studies have demonstrated that many patients experience a substantial degree of unrelieved pain following operative procedures and that this pain can increase the incidence of serious complications, the management of discomfort continues to be suboptimal. Narcotic analgesia is the mainstay of acute postoperative pain management but patient, clinician, and institutional barriers often limit the effectiveness of drug treatment. Furthermore, pharmacologic interventions alone may not address all the factors involved in the conscious experience of pain. Massage is a complementary or adjunctive medical technique that has been used for thousands of years. Yet there is scant research related to the use of massage therapy in postoperative pain management. Used in tandem with pharmacologic treatments, massage may have the potential to substantially improve acute pain relief.

OBJECTIVE(S):

The proposed research will test the hypotheses that: 1) perceived post-operative pain and anxiety decrease over time (5 days) more rapidly in the massage group compared with the focused attention and routine care groups; 2) perceived post-operative pain and anxiety are immediately reduced in the massage group compared with the focused attention and routine care groups. (differences in pre/post daily scores); 3) post-operative complication rate is reduced and function is improved by the adjuvant use of massage compared to the control groups; 4) the adjuvant use of massage reduces postoperative length of stay and cost of care; and 5) patient satisfaction with postoperative pain relief is enhanced by the adjuvant use of massage.

METHODS:

The study is a prospective, randomized clinical trial conducted at the Ann Arbor and Indianapolis VA medical centers. Patients undergoing operative procedures involving either a sternotomy or an abdominal incision at least 8 cm in length will be randomly assigned to one of three parallel treatment groups: 1) routine postoperative care, 2) focused attention where a massage therapist spends dedicated time (but no massage is given) with the patient once a day (20 min) during post-operative days 1 through 5; or 3) effleurage massage (20 min) performed by a massage therapist once per day on post-op days 1 through 5. The anticipated sample size is 582 patients. Postoperatively patients will be asked to rate their intensity of pain, well-being, function (ability to cough, deep breathe, sleep and activity level) daily for up to five days (less if discharged prior to day five). Data will be collected on all aspects of narcotic analgesia use including the name of each drug, dose, route, and time of administration. On day six patients will complete a survey to assess their satisfaction with pain management. Using the Department of Veterans Affairs National Surgical Quality Improvement Program (NSQIP) format, data will be collected on postoperative complications during the first 30 days after the procedure. Other factors relevant to the veteran population that may affect pain control will be assessed in relationship to pain management.

STATUS:

This study began in September 2002. We are currently in the data analysis phase of the project and plan to be finished by December, 2005.

IMPACT:

Although pharmacologic agents have the ability to effectively limit pain, acute postoperative pain is often poorly managed with analgesic drugs alone. This study will be the first large-scale randomized clinical trial of massage as a complementary treatment in the management of acute postoperative pain. This study will help to determine if massage can serve as a useful adjuvant therapy in the management of acute postoperative incisional pain. Results from this study would inform pain management guidelines and allow the VA and the scientific community to make informed decisions regarding the potential benefits of one form of CAM (Complimentary and Alternative Medicine).

ELIGIBILITY:
Inclusion Criteria:

Veterans undergoing major surgery with an incision that is greater than or equal to 8 cm in length

Exclusion Criteria:

Blindness, rash or skin lesions on the back, unable to read, florid psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-02; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Post-operative pain intensity and pain unpleasantness over 5 days post-surgery

SECONDARY OUTCOMES:
Anxiety, activity levels, function

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B. Hinshaw, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Dolores F. Cikrit, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States